CLINICAL TRIAL: NCT02150304
Title: Phase IV Study of Intravenous Aminophylline During Spinal Anesthesia
Brief Title: Aminophylline Prophylaxis For Postdural Puncture Headache
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İBRAHİM ÖZTÜRK, doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: PDPHAMINOPHYLLINE
Record Dates: First submitted 2014-05-24; First posted 2014-05-29 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- intravenous aminophylline: intravenous aminophylline use during spinal anesthesia
- no intravenous aminophylline: no use of intravenous aminophylline during spinal anesthesia

SUMMARY:
postdural puncture headache is a rare but serious complication of spinal anesthesia. many drugs were studied in prevention or treatment of that complication. However, there are limited numbers of trials about intravenous aminophylline for prevention. because of that we retrospectively aimed to investigate the effectiveness of aminophylline for postdural puncture headache in cesarean section.

DETAILED DESCRIPTION:
retrospective trial about the effect of intravenous aminophylline for prevention of PDPH after caserean section with spinal anesthesia

ELIGIBILITY:
Inclusion Criteria:

* patients aolder than 18 years old

Exclusion Criteria:

* conversion to general anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: patient records form who experinced headache after caserean section with spinal anesthesia were retrospectively evaluated
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
postdural puncture headache | postoperative 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim öztürk, M.D., Principal Investigator — dışkapı yıldırım beyazıt education and research hospital
Locations (1):
- Dışkapı Yıldırım Beyazıt Education and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Naghibi K, Hamidi M. Prophylactic administration of aminophylline plus dexamethasone reduces post-dural puncture headache better than using either drug alone in patients undergoing lower extremity surgery. Adv Biomed Res. 2014 Jan 9;3:5. doi: 10.4103/2277-9175.124631. eCollection 2014. PMID 24600595
- [Background] Basurto Ona X, Uriona Tuma SM, Martinez Garcia L, Sola I, Bonfill Cosp X. Drug therapy for preventing post-dural puncture headache. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD001792. doi: 10.1002/14651858.CD001792.pub3. PMID 23450533